CLINICAL TRIAL: NCT04795518
Title: The Pattern of Antibiotic Prescription for Children Among a Group of Pediatric Dentists.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed mostafa abdo elgendy, master degree student, Cairo University
Other Study IDs: antibiotic misues
Record Dates: First submitted 2021-03-05; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Antibiotic Resistant Strain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross sectional study by questionnaire among group of pediatric dentistry: An interviewed questionnaire is divided into two parts. The first part of the questionnaire will investigate the socio-demographic characteristics of the respondents. The second part of the questionnaire is divided into five sections to cover the following items:
  1. Use of antibiotics pattern
  2. Knowledge about antibiotics
  3. Sources of information

SUMMARY:
The aim of this study is to determine the pattern of antibiotic prescription for children among a group of pediatric dentists

DETAILED DESCRIPTION:
Antibiotic prescriptions for children is a cause for concern in both developed and developing countries, especially for its excessive use in non-established infections or in infections with viral etiology (Friedman et al., 2011). Although antibiotics play a crucial role in reducing child morbidity and mortality (De Jong et al., 2009), its irrational use directly increases antibiotic resistance by promoting the emergence of resistant bacteria leading to increased rates of treatment failures and more severe illness episodes with higher costs and mortality rates (Adisa et al., 2018).

Rational prescribing implies using the right drug for the right patient at the right time in the right dose and manner of administration at affordable cost with the right information. Thus, rational antibiotic prescription has to be tailor-made for individual patients taking into account the diagnosis, age, sex, weight, microorganism susceptibility, vital organ functions, drug and food interactions, as well as socioeconomic background of a patient (Aronson, 2014).

Within the dental community, awareness of clinical indications of antibiotic prescriptions to the child dental patient is lacking. It was found that a substantial proportion of children who received dental treatment for pain or localized swelling under general anaesthesia had also received antibiotics, with wide variation in antibiotic regimens (Dar-Odeh et al., 2018). Further, among members of the American Academy of Pediatric Dentistry, there was a trend toward overuse of antibiotics for non-indicated clinical conditions, like pain relief, irreversible pulpitis, and localized dentoalveolar abscess (Sivaraman et al., 2013).

Conditions requiring antibiotic treatment in dentistry is limited and there should be (i) a therapeutic goal to help treatment of acute/chronic infections (where drainage or debridement is impossible) or (ii) a prophylactic goal to prevent metastatic infections (e.g., bacterial endocarditis) or local or systemic spread of the infection (Dar-Odeh et al., 2010).

The non-clinical factors initiated antibiotic prescribing for some clinicians, such as unavailability of close appointments and seeking parental satisfaction (Sivaraman et al., 2013). A similar trend was observed in developing countries, where a substantial proportion of dentists prescribe for non-indicated clinical conditions, such as dry socket, localized periapical infection, marginal gingivitis, periodontitis, and pulpitis (Kouidhi et al., 2011). This insufficient knowledge of the appropriate clinical indications is paralleled by a lack of awareness of important interventions that promote the optimal use of antibiotics, such as antibiotic stewardship programs. Other forms of abuse in prescribing antibiotics include prescribing broad-spectrum antibiotics for infections that can be treated by narrow-spectrum antibiotics, prescribing antibiotics for long periods, and adopting inappropriate dosing regimens (Sivaraman et al., 2013).

Patients who consult their GP due to tooth-related problems are unlikely to receive a surgical intervention and have a greater likelihood of being prescribed a systemic antibiotic compared to individuals who consult a dentist with similar symptoms (Cope et al., 2015)complications from an odontogenic infection, (Seppänen et al., 2011) the management of dental problems in general practice could result in increased patient morbidity. Furthermore, the indiscriminate use of antibiotics may contribute to the emergence of antibiotic-resistant bacterial strains (Cope et al., 2015).

Antibiotic resistance (AR) is a condition when bacteria change against antibiotics which are developed to cure the illnesses they cause. It is a global crisis and posed as one of the greatest threats to population health. This problem is driven by many factors such as low quality of antibiotics and improper (under- or over-) use of antibiotics (including self-medication) (Alumran et al., 2013). Self-medication, which refers to the use of any medical products without a prescription or following unprofessional recommendations in treating any illnesses (Togoobaatar et al., 2010), is particularly leading to the AR. Self-medication practice possibly raises incorrect drug selection, drug resistance, uncontrolled adverse effects or drug reactions, misdiagnosis, and delay in medical care (El-Hawy et al., 2017).

It has been observed that contribute to the problem of antibiotic resistance by dentists can be substantial as dentists prescribe 10% of all common antibiotics. Yingling et al concluded from the findings of his study among members of the American Association of Endodontists (AAE) that they were prescribing antibiotics inappropriately. On the contrary (Yingling et al., 2002), the National Center for Disease Control and Prevention found that almost one-third of all outpatient antibiotic prescriptions are unnecessary (Swift and Gulden, 2002). The world has entered an era where some bacterial species are resistant to the full range of antibiotics presently available, with the methicillin-resistant Staphylococcus aureus and vancomycin-resistant Staphylococcus aureus being the most widely known example of extensive resistance (Lewis, 2008).

It is estimated that, in 2050, there will be more than 10 million deaths and 100 trillion USD lost due to AR if no substantial actions have been made to eliminate this emerging threat. As inappropriate antibiotic use is the primary cause of AR, responses to this phenomenon prioritize promoting public awareness about AR (El-Hawy et al., 2017).

Irrational prescribing can be due to errors such as required amount of drug or as errors in writing, abbreviations, pharmaceutical form, drug dosage, administration method, or duration of treatment. These errors can lead to ineffective treatment and dangerous, long-lasting illness, or worse: harm to the patient and an increase of the cost of treatment (Grant et al., 2013).

Dentists, like other health care practitioners should have sufficient knowledge about drugs. Observing the prescription principles according to international law for dentists is required. Although dental prescription generally contain pharmaceutics items are limited to providing short-term drug therapy or specific drugs prescribed for dental surgeries but the evidence suggests that in many countries, dentists often do not enjoy a good medical knowledge for this reason, some mistakes in writing prescription occurred (Guzmán-Álvarez et al., 2012).

Goud et al. reported that general dentists prescribed more than required antibiotics for root canal therapy (Goud et al., 2012). Mendonca et al. found that in one-fourth of prescriptions written by dentists, medication names were illegible (Mendonça et al., 2010). Ogunbodede et al findings indicate the presence of different types of error in dentist's prescription in term of dosing, frequency and duration of drug use (Ogunbodede et al., 2005).

ELIGIBILITY:
Inclusion Criteria:

Dentists of pediatric dentistry working for children aged. Dentists who have BDS degree in the last 20 years.

Exclusion Criteria:

-

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Group of pediatric dentists
Sampling Method: Probability Sample
Enrollment: 334 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Pattern of antibiotic prescription in children | baseline
  Questionnaire (Kaul et al., 2018), Multiple choice question

CONTACTS AND LOCATIONS:
Overall Officials: ahmed M EL-Gendy, BDS, Principal Investigator — Dentist at Ministry of Health,EGYPT; Fatma Kl EL-Gendy, PhD, Study Chair — Assistant Professor at Pediatric Dentistry and Dental Public Health Department
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

REFERENCES:
- [Result] Kaul R, Angrish P, Jain P, Saha S, V Sengupta A, Mukherjee S. A Survey on the Use of Antibiotics among the Dentists of Kolkata, West Bengal, India. Int J Clin Pediatr Dent. 2018 Mar-Apr;11(2):122-127. doi: 10.5005/jp-journals-10005-1497. Epub 2018 Apr 1. PMID 29991865